CLINICAL TRIAL: NCT05685498
Title: Peer-led HIV Self-testing to Improve HIV Testing and Linkage to HIV Care Among Men in Two Fishing Communities in Rural Uganda: a Pilot Intervention
Brief Title: Peer-led HIV Self-testing Among Men in Two Ugandan Fishing Communities
Acronym: PEST4MEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joseph KB Matovu (Other)
Collaborators: Makerere University (Other); RAND (Other)
Responsible Party: Sponsor-Investigator, Joseph KB Matovu, Senior Lecturer, Busitema University
Organization: Busitema University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BusitemaU
Record Dates: First submitted 2022-12-21; First posted 2023-01-17 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: HIV Testing
Keywords: HIV self-testing; Men; Fishing communities; Uganda
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer-led HIV self-testing among male fisherfolk in Uganda (Other): Men aged 15 years or older, who self-report a HIV-negative or unknown HIV status at enrolment and last tested for HIV three or more months are enrolled into the study. Enrolled men receive two HIV self-test kits from a trained community-based distributor (or peer-leader). Peer-leaders are selected from existing social networks and are trained in HIV self-testing procedures prior to distributing HIV self-test kits. The goal of the study is to assess if distribution of HIV self-test kits to men through trained local peer-leaders is feasible and acceptable in a fishing community context, and whether this approach can help to improve access to HIV testing services and, by implication, improve HIV testing uptake and subsequent linkage to appropriate HIV prevention, care and treatment services. Men are interviewed at baseline will be followed up at 1, 6 and 12 months post-baseline to determine HIV testing uptake, linkage to and retention in HIV care.
  Interventions: Behavioral: Peer-led HIV self-testing among male fisherfolk in Uganda

INTERVENTIONS:
Behavioral: Peer-led HIV self-testing among male fisherfolk in Uganda — This behavioral intervention is centered on the distribution of HIV self-test kits to men through their respective peer-leaders. The investigators have identified up to 18 social network groups; each group is represented by 1-2 peer-leaders who were selected during community engagement meetings. Peer-leaders have received a 3-day training in the HIV self-testing processes, communication skills, existing referral mechanisms, and basic counseling skills. After the training, each peer-leader nominated up to 20 male members (15+ years) from within their social networks who were screened for study eligibility. Eligible male social network members were administered a baseline interview and requested to go to their peer-leaders to obtain their HIV self-test kits.

SUMMARY:
The goal of this behavioral interventional study is to assess the feasibility and acceptability of a peer-led HIV self-testing intervention among men in two fishing communities along the shores of Lake Victoria in Uganda. The main objectives of the study are: a) to assess the feasibility of implementing a peer-led HIV self-testing intervention among men in a fishing community context; b) determine the uptake of HIV self-testing among men in the fishing communities, and c) determine linkage to and retention in HIV care among newly diagnosed HIV-positive men following peer-led HIV self-testing. Participants will:

* Be administered a baseline questionnaire to assess prior HIV testing behaviors and willingness to self-test for HIV
* Receive two HIV self-test kits, one for them and one for someone else that they prefer to give the kit, to determine HIV testing behaviors among men and their significant others
* Be administered follow-up questionnaires at one (1), six (6) and 12 months post-baseline to determine linkage to and retention in HIV care among those testing HIV-positive, as well as linkage to appropriate HIV prevention services among those testing HIV-negative.

DETAILED DESCRIPTION:
Background

In this study, investigators propose to use a social network-based, peer-led HIV self-testing model to assess uptake of HIV testing, as well as linkage to appropriate HIV prevention, care and treatment services in two high HIV prevalence island districts with limited access to HIV and other health services.

Primary aims

1. Compare approaches for peer-leader selection in two fishing communities in order to identify suitable peer-leader selection approaches for typical fishing communities.
2. Assess uptake of HIV testing services associated with peer-led HIV self-testing among men living in two high HIV prevalence fishing communities
3. Assess the effect of a peer-led HIV self-testing (HIVST) model in: (i) identifying previously undiagnosed HIV infections; (ii) improving linkage to HIV care among newly identified HIV-positive individuals; and (iii) improving retention in HIV care among linked HIV-positive individuals

Study sites The intervention will be conducted in two different fishing communities (one in each district) located in two high HIV prevalence island districts of Buvuma and Kalangala, located in Lake Victoria, Uganda.

Intervention Description The peer-led HIV self-testing intervention will include distribution of HIV self-test kits through trained male peer-leaders. Forty peer-leaders will be selected through community meetings held in each fishing community. The following sub-sections describe the key components of the intervention.

1. Training of selected peer-leaders and distribution of HIV self-test kits Selected peer-leaders will be trained in HIV self-testing processes and procedures for a period of three days after which they will be asked to nominate up to 20 male members (15+ years) from their social network. All the nominated social network members will be screened for eligibility and up to 400 eligible men will be enrolled into the study. Peer-leaders will receive the number of kits equal to the number of eligible members enrolled from their social network for up to 20 kits per peer-leader. Peer-leaders will receive a one-time facilitation allowance to facilitate their movement in the community during the process of distributing HIV self-test kits to members of their social network. As part of the distribution process, peer-leaders will be requested to demonstrate to their social network members how the HIV self-testing process is done, including how to obtain the oral swab, how to time the 20 minutes needed for the kit to show results, and how to read and interpret results.
2. Antiretroviral therapy initiation through health facility-coordinated mobile outreaches Given that fishing communities do not usually have health facilities within their proximity, many HIV-positive individuals tend to miss conventional HIV testing and linkage to HIV care services. To address this gap, investigators intend to work with mainland health facilities nearest to the targeted fishing communities to conduct health outreach sessions in which HIV testing and linkage to HIV will be provided as part of a multi-disease health promotional campaign. Study participants will be notified through their peer-leaders regarding when the health outreach sessions will be conducted and they will be requested to come and access free health services, including confirmatory HIV testing. Study participants who will be confirmed as HIV-positive will be provided with an initial dose of antiretroviral therapy (at the same outreach session) lasting until the next outreach session or until they are linked to an existing community client-led ART delivery (CCLAD) group, while those confirmed as HIV-negative will be linked to appropriate HIV prevention services including condom promotion and male circumcision services, as appropriate.
3. Peer-facilitated retention in HIV care Retention in HIV care is an ongoing challenge in HIV care and treatment programs. At the time of linkage to HIV care, the investigators will ask HIV-positive individuals if they have anyone within their close network that can act as their treatment buddy (including their peer-leader); someone who could help to pick their drugs at the planned outreach sessions in the event that they cannot do so, or provide them with psycho-social support as needed in order to help them continue to take their HIV treatment as recommended. If they agree, social network members will be asked if they have ever disclosed their HIV positive status to that person, and if not, they will be asked if they would like to disclose to them on their own or whether they would need to be assisted to accomplish the HIV status disclosure process. The investigators will explore if disclosure to a peer-leader (as opposed to someone else within the network) facilitates retention in HIV care.

Data collection procedures and methods

Data will be collected through two inter-related phases: In phase 1, the investigators will collect qualitative data (through focus group discussions) on men's perception of HIV self-testing as an HIV testing strategy as well as their perceptions on receiving HIV self-test kits from trained male peer-leaders who are members of their community. Focus group discussions (FGDs) will be composed of between 8 and 12 men. Investigators will conduct six FGDs to explore people's perceptions on oral HIVST, strategies that can be used to distribute HIVST kits to men in a fishing community; and qualities of men that can be selected as peer-leaders, among other aspects. Because investigators intend to ask peer-leaders to facilitate linkage to HIV care among men who test HIV-positive, investigators will also seek people's perceptions about the acceptability of peer-leaders knowing people's status and helping with linkage to care. FGDs will be conducted by trained interviewers with experience in the conduct of qualitative interviews. All FGDs will be audio-recorded (with permission from the participants) and transcribed verbatim by the same interviewers that will have collected the data.

In phase 2, investigators will collect baseline and follow-up data necessary to assess the acceptability of a peer-led HIVST intervention as well as linkage to appropriate HIV prevention, care and treatment services, and retention in HIV care among HIV-positive social network members. This phase will be implemented through four inter-related steps:

Step 1 (Screening for eligibility): All social network members recommended to the study will be screened for eligibility to participate in the study using a screening tool. Only individuals recommended by peer-leaders (who will also appear on a peer-leader's pre-generated list) will be screened for eligibility, and those found to be eligible will be enrolled into the study.

Step 2 (Baseline interview): All eligible social network members will be administered a baseline interview to collect socio-demographic and behavioural data, as well as data on participants' willingness to receive HIVST kits from peer-leaders, and their willingness to disclose their HIV status to a peer-leader on their own volition. Data will be collected by trained interviewers with experience in the conduct of quantitative interviews. Participants will receive a travel refund and compensation for time after participating in the baseline interviews. The baseline findings will provide the study team with information needed to measure the success or failure of the intervention.

Step 3 (Follow-up visits): Follow-up interviews will be conducted at 1, 6 and 12 months post-baseline, using a follow-up questionnaire uploaded on open-data kit-enabled phones. During follow-up, individuals who received HIVST kits will be asked whether or not they used them to test for HIV. Those that will have failed to use the kits will be asked in open-ended questions to state reasons for their failure while those that will have used the kits will be asked about HIVST experiences (both positive and negative). Investigators will assess if individuals who self-tested for HIV sought confirmatory HIV testing, and if they did, whether or not they received their HIV test results. Individuals who will link to HIV care will be followed up to determine if they are still in HIV care at 6 and 12 months post-baseline. Individuals who will report that they tested HIV-positive but were yet to link to HIV care will be asked about the reasons for the delay and whether they plan to link to care in the future.

Step 4 (Post-intervention qualitative interviews): At the end of the study (i.e. after month-12 follow-up visit), qualitative data will be collected from all the peer-leaders to document process issues around the distribution of HIVST kits and suggestions on how best the HIVST distribution process can be improved in the future. Investigators will conduct in-depth interviews with 30 men. Qualitative data will be collected using key informant and in-depth interview guides after obtaining written, informed consent from the participants.

ELIGIBILITY:
Inclusion Criteria:

* Age 15 years or older
* Residence in the targeted fishing community (and intended to stay for 12 or more months)
* Self-reported HIV-negative or unknown HIV status at enrolment
* Last HIV test was done three or more months from the time of enrolment

Exclusion Criteria:

* Men reporting a history of intimate partner violence in the past year preceding the survey
* Men who did not belong to pre-identified social networks in the community
* Men who were mentally incapacitated to understand the informed consent process
* Unemancipated minors aged 15-17 years

Min Age: 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of men who have self-tested for HIV | One month from the time of receiving the kits.
  Men will receive HIV self-test kits and be trained in how to use them as well as read and interpret results by trained peer-leaders. Uptake of HIV self-testing will be defined as the percentage of those that received HIV self-test kits from their peer-leaders who actually used them to self-test for HIV.
Percentage of men with confirmed HIV-positive results who have been linked to HIV care | One to six months after a HIV-positive self-test result
  As per the manufacturer's instructions, all men with HIV-positive self-test results will be required to seek confirmatory HIV testing at the nearest health facility or at an outreach event, as case may be. For this outcome, we will aim to assess the percentage of men with confirmed HIV-positive results who have been linked to HIV care services (i.e. the percentage of men with confirmed HIV-positive results who have been started on antiretroviral therapy as per Uganda's national test and treat policy).
Percentage of linked HIV-positive men who have been retained in HIV care | Six to 12 months after linkage to HIV care
  Investigators will aim to assess the percentage of linked HIV-positive results who have been retained in HIV care (i.e. percentage of linked HIV-positive men who will still be receiving their antiretroviral therapy over the study duration).

SECONDARY OUTCOMES:
Percentage of men with confirmed HIV-positive results who have disclosed their HIV-positive status to their peer-leaders | Six to 12 months after HIV self-testing
  Investigators will determine the percentage of men with confirmed HIV-positive results who have disclosed their HIV sero-positive status to their peer-leaders. This will help us to determine if disclosure to a peer-leader can improve linkage to HIV care among HIV-positive men.
Percentage of men with confirmed HIV-positive results who have been linked to HIV care at community-based mobile outreaches. | Six to 12 months after HIV self-testing
  Investigators will assess if mobile outreaches conducted in conjunction with the nearest health facilities can improve linkage to HIV care among HIV-positive men living in isolated fishing communities with limited access to HIV and other health services.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph KB Matovu, PhD, Principal Investigator — Busitema University
Locations (2):
- Uganda (2):
  - Buvuma district, Buikwe
  - Kalangala District, Kalangala

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data will be available to other users, including students who are pursuing their graduate studies at Busitema University and junior faculty but no individual participant data sharing plans have been finalized at the moment. Students and junior faculty will have access to HIV testing and linkage to HIV care data, and to any other data collected as part of this study, after the primary and secondary objectives of this study have been addressed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 24 months after the end of the last follow-up visit.
Access Criteria: Individual data users will be required to submit a request to the study PI by email indicating the primary question that they intend to answer and the type of data that they need. After a careful review of the request received, de-identified individual data will be availed to the person requesting the data. While data will be generally available to researchers with or without Busitema University Faculty of Health Sciences, only students enrolled at Busitema University Faculty of Health Sciences or Makerere University School of Public Health will have access to the data.

REFERENCES:
- [Derived] Matovu JK, Namwama AT, Kemigisha L, Taasi G, Nakabugo J, Wandabwa J, Bogart LM, Fakier N, Wanyenze RK, Olupot-Olupot P, Musinguzi J, Serwadda D. Feasibility, acceptability and preliminary effects of a social network-based, peer-led HIV self-testing intervention among men in two Ugandan fishing communities, 2022. Arch Public Health. 2025 Jan 24;83(1):23. doi: 10.1186/s13690-025-01511-9. PMID 39849572